CLINICAL TRIAL: NCT07140614
Title: A First-in-human, Multi-center, Randomized, Participant- and Investigator-blinded, Placebo Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of EDK060 in Adults With Charcot-Marie Tooth Type 1A (CMT1A).
Brief Title: A First in Human Study to Assess the Safety, Tolerability, and Pharmacokinetics of EDK060 in Adults With CMT1A.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEDK060A12101
Record Dates: First submitted 2025-08-22; First posted 2025-08-24 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Charcot-Marie-Tooth Disease, Type 1A
Keywords: CMT1A
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EDK060 (Experimental): Doses A; B; C; D
  Interventions: Drug: EDK060, dose A; Drug: EDK060, dose B; Drug: EDK060, dose C; Drug: EDK060, dose D
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: EDK060, dose A — EDK060, dose A, Single dose, IV infusion
  Arms: EDK060
Drug: EDK060, dose B — EDK060, dose B, Single dose, IV infusion
  Arms: EDK060
Drug: EDK060, dose C — EDK060, dose C, Single dose, IV infusion
  Arms: EDK060
Drug: EDK060, dose D — EDK060, dose D, Single dose, IV infusion
  Arms: EDK060
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to characterize the safety, tolerability, and pharmacokinetics of EDK060 as compared to placebo in adult patients with CMT1A.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent before any assessment is performed.
* Be male or female and 18 to 60 (inclusive) years of age at the time of screening.
* Participant must have a clinical diagnosis of Charcot-Marie-Tooth Disease Type 1A (CMT1A) including verified documentation of genetic testing showing duplication of the PMP22 gene by an accredited/certified laboratory (according to local regulations)
* Have detectable upper extremity nerve conduction velocities (sensory and motor) in at least one extremity at screening.

Exclusion Criteria

* Unable to communicate well with the investigator, to understand and comply with the visits and procedures of the study.
* History of cardiac, renal, liver, hematological, immune system disorders.
* Pregnant/nursing female participants. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for the duration of the follow-up period. Sexually active males unless they use a condom during intercourse.
* Inability or unwillingness to provide serial skin biopsy samples.
* Inability or unwillingness to undergo repeated venipuncture or in the opinion of the investigator, participant would be at an increased risk for adverse events related to these procedures.
* Use of any drug intended to modify the course of CMT1A within 6 months from screening, including but not limited to: PTX-3003 (baclofen, sorbitol, and naltrexone in combination).
* History of compression neuropathy within the last 6 months from screening and/or other conditions that can cause peripheral neuropathy, including but not limited to diabetes, chronic alcoholism, exposure to neurotoxic medications, exposure to environmental neurotoxins, traumatic nerve injury, thyroid disease, or infections.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2028-02-25 (Estimated); Study Completion 2028-02-26 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From baseline up to day 140
  Incidence of AEs and SAEs by treatment group, including changes in vital signs, laboratory measures, neurological examinations and electrophysiology measures qualifying and reported as AEs.

SECONDARY OUTCOMES:
EDK060 Plasma PK parameters - Cmax | From baseline up to day 140
  The maximum (peak) observed EDK060 plasma concentration after single dose administration (mass x volume-1)
EDK060 Plasma PK parameters - Tmax | From baseline up to day 140
  The time to reach maximum (peak) plasma, EDK060 concentration after single dose administration (time)
EDK060 Plasma PK parameters - AUClast | From baseline up to day 140
  The area under the concentration-time curve of EDK060 from time zero to the last measurable concentration sampling time (tlast) (mass x time x volume-1)

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Novartis Investigative Site, Ottawa, Ontario
  - Montreal Neurological Institute, Montreal, Quebec
  - CIUSS de l´Estrie-CHUS- Hôpital Fleurimont, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No